CLINICAL TRIAL: NCT04468438
Title: Role of Estrogen in the Flarring up of Lupus Nepheritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager Zanaty Abdelraouf, Principal investigator, Assiut University
Other Study IDs: Example 3
Record Dates: First submitted 2020-01-29; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2019-11

CONDITIONS: Activity of Lupus Nepheritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 50 patients with LN with regular menstrual cycle: 1- First group of50 patients with regular menstrual cycle
  Interventions: Diagnostic Test: serum estrogen and urinary albumin creatinine ratio
- 50 patients with LN with amenorrhea: 2- Second group of 50 patients with amenorrhea.
  Interventions: Diagnostic Test: serum estrogen and urinary albumin creatinine ratio

INTERVENTIONS:
Diagnostic Test: serum estrogen and urinary albumin creatinine ratio — serum estrogen and urinary albumin creatinine ratio

SUMMARY:
Role of estrogen in the flarring up of lupus nepheritis

DETAILED DESCRIPTION:
Systemic lupus erythematosus SLE is an autoimmune disease that affects ∼5.5 per 100,000 individuals worldwide . SLE is characterized by loss of tolerance against nuclear autoantigens, lymphoproliferation, polyclonal autoantibody production, immune complex disease, and multiorgan tissue inﬂammation. Up to 50% of SLE patients develop some degree of renal involvement, with up to 20% progressing to end-stage renal disease, depending on racial background . Lupus nephritis LN is characterized by anti-nuclear Ab production, immune complex deposition, and immune-mediated kidney damage. Development of LN remains a sign of poor prognosis and is a signiﬁcant cause of morbidity and mortality . Because 9 of 10 SLE patients are women, the role of the sex hormones estrogens in this disease is of key interest. Estrogens signal through two receptors: estrogen receptor a ERa and estrogen receptor b ERb. In contrast to estrogen receptor b, ERa is found in female reproductive organs, yet is robustly expressed in kidney, liver, heart, and lungs in males and females,as well as on most immune cells however the kidney is considered the most estrogenic nonreproductive organ. The overwhelming female predominance for SLE begins at puberty and extends to menopause , supporting the concept that estrogens or other reproductive factors stimulate lupus development. This concept is further evidenced by reports of menstrual cycle flares of SLE , disease exacerbations by oral contraceptives or estrogen administration , and induction of lupus by ovulation regimens . Ultraviolet rays has arole in the flarring up SLE. There is evidence that fibroblasts and blood lymphocytes from SLE patients are hypersensitive to the cytotoxic effects of UV light radiation

. RNA and protein synthesis is also affected by UV light 18. A study from 1986 found that people were more likely to menstruate during a new moon, which occurs during the opposite half of the lunar cycle than the full moon . There are different evolutionary theories speculating why the human menstrual cycle length evolved to be so close to the lunar cycle in length. Stories and beliefs connecting the two are also found in various cultures and mythologies . The terms menstruation and menses even come from Latin and Greek words meaning month mensis and moon mene

ELIGIBILITY:
Inclusion Criteria:

1. Patients with SLE complicated with LN.
2. Patients with age more than 18 years old.

Exclusion Criteria:

* 1- Pragnancy, lactation. 2- Menpause. 3- Primary amenorrhea. 4- Patients with current use of oral contraceptive agents. 5- Patients who receive pulse therapy during the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female patients at the reproductive age with systemic lupus
Study Population: female patients at the reproductive age with systemic lupus divided into two groups:
  1. First group patients with regular menstrual cycle.
  2. Second group patients with amenorrhea.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Role af estrogen in flarring up of lupus nepheritis to detect time of pulse therapy | one year
  Measurement of estrogen in the first day of menstruation and the14th day of menstruation To intensify treatment during days of menstruation or days of full moon.

REFERENCES:
- [Background] Somers EC, Marder W, Cagnoli P, Lewis EE, DeGuire P, Gordon C, Helmick CG, Wang L, Wing JJ, Dhar JP, Leisen J, Shaltis D, McCune WJ. Population-based incidence and prevalence of systemic lupus erythematosus: the Michigan Lupus Epidemiology and Surveillance program. Arthritis Rheumatol. 2014 Feb;66(2):369-78. doi: 10.1002/art.38238. PMID 24504809
- [Background] Tan DA, Haththotuwa R, Fraser IS. Cultural aspects and mythologies surrounding menstruation and abnormal uterine bleeding. Best Pract Res Clin Obstet Gynaecol. 2017 Apr;40:121-133. doi: 10.1016/j.bpobgyn.2016.09.015. Epub 2016 Oct 26. PMID 27863914
- [Background] Liu Z, Davidson A. Taming lupus-a new understanding of pathogenesis is leading to clinical advances. Nat Med. 2012 Jun 6;18(6):871-82. doi: 10.1038/nm.2752. PMID 22674006
- [Background] Moulton VR, Tsokos GC. Abnormalities of T cell signaling in systemic lupus erythematosus. Arthritis Res Ther. 2011 Mar 17;13(2):207. doi: 10.1186/ar3251. PMID 21457530